CLINICAL TRIAL: NCT05127486
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Galcanezumab Versus Rimegepant in Adult Participants With Episodic Migraine
Brief Title: A Study of Galcanezumab (LY2951742) in Adult Participants With Episodic Migraine
Acronym: CHALLENGE-MIG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18256; I5Q-MC-CGBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-11-03; First posted 2021-11-19 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Migraine; Episodic Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — galcanezumab; rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Galcanezumab (Experimental): Participants received a loading dose of 2 injections of 120 milligrams (mg) galcanezumab subcutaneously (SC) in the first month followed by 120 mg monthly for remaining 2 months.
  1 placebo oral disintegrating tablet (ODT) every other day for 3 months was given to preserve blinding.
  Interventions: Drug: Galcanezumab; Drug: Placebo
- Rimegepant (Active Comparator): Participants received 75 mg Rimegepant oral disintegrating tablet (ODT) every other day for 3 months.
  2 placebo SC injections loading dose, then 1 placebo SC injection monthly for remaining 2 months was given to preserve blinding.
  Interventions: Drug: Rimegepant; Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SC.
  Other Names: LY2951742
  Arms: Galcanezumab
Drug: Rimegepant — Administered orally.
  Arms: Rimegepant
Drug: Placebo — Administered orally.
  Arms: Galcanezumab
Drug: Placebo — Administered SC.
  Arms: Rimegepant

SUMMARY:
The purpose of this study is to assess whether galcanezumab is superior to rimegepant in the prevention of migraine in participants with episodic migraine. The study duration will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine, with or without aura, as determined by the study investigator and in consideration of International Headache Society International Classification of Headache Disorders - 3rd edition guidelines (ICHD-3 2018)

Exclusion Criteria:

* Have a known hypersensitivity to rimegepant or galcanezumab, and their excipients, monoclonal antibodies or other therapeutic proteins
* Have acute cardiovascular events and/or serious cardiovascular risk, or have had myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft, or stroke within 6 months of screening, or have planned cardiovascular surgery or percutaneous coronary angioplasty.
* Evidence of significant psychiatric disease by medical history, such as schizophrenia, personality disorders, or other serious mood or anxiety disorders.
* Women who are pregnant or nursing
* Current use or prior exposure to any calcitonin gene related peptide (CGRP) antagonist (small molecule or antibody) for any indication, including those who have previously completed or withdrawn from this study or any other study investigating a CGRP antagonist (small molecule or antibody)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (76):
- United States (76):
  - Gilbert Neurology, Gilbert, Arizona
  - Foothills Research Center / CCT Research, Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC Tempe, Tempe, Arizona
  - Velocity Clinical Research, Banning, Banning, California
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - Wr- Pri, Llc, Encino, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - California Medical Clinic for Headache and The Los Angeles Headache Center (Research Facility), Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Anderson Clinical Research, Redlands, California
  - Center for Clinical Trials of Sacramento, Sacramento, California
  - Velocity Clinical Research, Huntington Park, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Innovative Research of West Florida, Clearwater, Florida
  - AMR Miami, Coral Gables, Florida
  - Accel Research Sites- Clinical Research Unit, DeLand, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Accel Research Sites-LKD CRU, Lakeland, Florida
  - Visionary Investigators Network, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - University of South Florida, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - DelRicht Research, Atlanta, Georgia
  - Better Health Clinical Research, Newnan, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Chicago Headache Center, Chicago, Illinois
  - American Health Network of Indiana, LLC - Avon, Avon, Indiana
  - Deaconess Clinic, Evansville, Indiana
  - Alliance for Multispecialty Research, LLC El Dorado, El Dorado, Kansas
  - Alliance for Multispecialty Research, LLC Lexington, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - DelRicht Research, Covington, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - MedPharmics, LLC, Gulfport, Mississippi
  - Healthcare Research Network - St. Louis, Hazelwood, Missouri
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurosciences Research Center (Research Facility), Amherst, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Tekton Research, Edmond, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - DelRicht Research, Tulsa, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Velocity Clinical Research, Grants Pass (Research Facility), Grants Pass, Oregon
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Premier Neurology Research, P.C., Greer, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Tekton Research (Research Facility), Austin, Texas
  - FutureSearch Trials of Neurology, Austin, Texas
  - ACRC Trials, Austin, Texas
  - ACRC Trials, Carrollton, Texas
  - Velocity Clinical Research, Austin, Cedar Park, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Accurate Clinical Management - Houston, Houston, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Humble, Texas
  - Ventavia Research Group - Keller, Keller, Texas
  - ACRC Trials, Plano, Texas
  - Alpine Research Organization, Clinton, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Alliance for Multispecialty Research, LLC - AMR Norfolk, Norfolk, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Background] Schwedt TJ, Myers Oakes TM, Martinez JM, Vargas BB, Pandey H, Pearlman EM, Richardson DR, Varnado OJ, Cobas Meyer M, Goadsby PJ. Comparing the Efficacy and Safety of Galcanezumab Versus Rimegepant for Prevention of Episodic Migraine: Results from a Randomized, Controlled Clinical Trial. Neurol Ther. 2024 Feb;13(1):85-105. doi: 10.1007/s40120-023-00562-w. Epub 2023 Nov 10. PMID 37948006
- See also: A Study of Galcanezumab (LY2951742) in Adult Participants With Episodic Migraine (CHALLENGE-MIG) — https://trials.lillytrialguide.com/en-US/trial/muhFfaGNSBYar2xzfLSZR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Galcanezumab | Rimegepant
Started | 287 | 293
Received at Least 1 Dose of the Study Drug | 287 | 293
Completed | 261 | 266
Not Completed | 26 | 27
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Physician Decision | 4 | 1
Not completed — Withdrawal by Subject | 14 | 13
Not completed — Lost to Follow-up | 5 | 8

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Galcanezumab: Participants received a loading dose of 2 injections of 120 mg galcanezumab SC in the first month followed by 120 mg monthly for remaining 2 months.
  1 placebo ODT every other day for 3 months was given to preserve blinding.
- Rimegepant: Participants received 75 mg Rimegepant ODT every other day for 3 months.
  2 placebo SC injections loading dose, then 1 placebo SC injection monthly for remaining 2 months was given to preserve blinding.
- Total: Total of all reporting groups
Arm/Group | Galcanezumab | Rimegepant | Total
Number analyzed (Participants) | 287 | 293 | 580
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (12.6) | 42.3 (11.32) | 42.0 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 238 | 482
  Male | 43 | 55 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 65 | 131
  Not Hispanic or Latino | 219 | 223 | 442
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 8 | 11 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 34 | 44 | 78
  White | 236 | 232 | 468
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 287 | 293 | 580
Number of Monthly Migraine Headache Days [Mean (Standard Deviation); unit: days per month] — A Migraine Headache Day is defined as a calendar day on which a migraine headache or probable migraine headache occurred.
  days per month | 8.5 (2.85) | 8.3 (2.92) | 8.4 (2.89)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 50% Response Rate Across the 3-month Treatment Period.
Description: A migraine headache day is a calendar day on which a migraine headache or probable migraine headache occurred. Overall mean percentage across months 1 through 3 of participants with at least a 50% reduction in monthly migraine headache days from baseline (50% response rate) using a categorical pseudo likelihood-based repeated measures model for binary responder indicator with fixed, categorical effects of treatment, month, treatment by month, and continuous, fixed covariate of baseline monthly migraine headache day.
Time Frame: Baseline, Month 1 through Month 3
Population: All randomized participants who received at least one dose of study drug and had non-missing baseline value and at least one non-missing post-baseline value for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 269 | 284
percentage of participants | 62 | 61
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Test type: Superiority; p = 0.695, pseudo likelihood-based repeated measure; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.81 to 1.38]

2. Secondary Outcome: Percentage of Participants With 75% Response Rate Across the 3-month Treatment Period.
Description: A migraine headache day is a calendar day on which a migraine headache or probable migraine headache occurred. Overall mean percentage across months 1 through 3 of participants with at least a 75% reduction in monthly migraine headache days from baseline (75% response rate) using a categorical pseudo likelihood-based repeated measures model for binary responder indicator with fixed, categorical effects of treatment, month, treatment by month, and continuous, fixed covariate of baseline monthly migraine headache day.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 269 | 284
percentage of participants | 37 | 33
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Test type: Superiority; pseudo likelihood-based repeated measure; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.89 to 1.56]

3. Secondary Outcome: Percentage of Participants With 100% Response Rate Across the 3-month Treatment Period.
Description: A migraine headache day is a calendar day on which a migraine headache or probable migraine headache occurred. Overall mean percentage across months 1 through 3 of participants with at least a 100% reduction in monthly migraine headache days from baseline (100% response rate) using a categorical pseudo likelihood-based repeated measures model for binary responder indicator with fixed, categorical effects of treatment, month, treatment by month, and continuous, fixed covariate of baseline monthly migraine headache day.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 269 | 284
percentage of participants | 18 | 15
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Test type: Superiority; pseudo likelihood-based repeated measure; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.89 to 1.79]

4. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days Across the 3-month Treatment Period.
Description: A migraine headache day is a calendar day on which a migraine headache or probable migraine headache occurred. Overall mean was derived from the average of month 1 through month 3. Least square (LS) mean was calculated using mixed model for repeated measures (MMRM) model with treatment, month, and treatment-by-month interaction as fixed effects and baseline number of migraine headache days, and baseline-by-month interaction as continuous variables.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days per month
Groups:
- 75 mg Rimegepant: Participants received 75 mg Rimegepant ODT every other day for 3 months.
  2 placebo SC injections loading dose, then 1 placebo SC injection monthly for remaining 2 months was given to preserve blinding.
Arm/Group | Galcanezumab | 75 mg Rimegepant
Number analyzed (Participants) | 269 | 284
days per month | -4.75 (0.17) | -4.39 (0.16)
Statistical Analysis 1: Comparison: Galcanezumab vs 75 mg Rimegepant; Test type: Superiority; Mixed Models Analysis; LS Mean difference = -0.37, 95% CI 2-sided [-0.82 to 0.09]

5. Secondary Outcome: Mean Change From Baseline in the Number of Monthly Migraine Headache Days at Month 1
Description: A migraine headache day is a calendar day on which a migraine headache or probable migraine headache occurred. LS mean was calculated using MMRM model with treatment, month, and treatment-by-month interaction as fixed effects and baseline number of migraine headache days, and baseline-by-month interaction as continuous variables.
Time Frame: Baseline, Month 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days per month
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 266 | 275
days per month | -4.33 (0.20) | -3.77 (0.20)
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Test type: Superiority; Mixed Models Analysis; LS Mean difference = -0.55, 95% CI 2-sided [-1.11 to 0.00]

6. Secondary Outcome: Mean Change From Baseline in the Number of Monthly Migraine Headache Days at Month 2
Description: as for outcome 5
Time Frame: Baseline, Month 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days per month
Arm/Group | Galcanezumab | 75 mg Rimegepant
Number analyzed (Participants) | 256 | 268
days per month | -4.81 (0.20) | -4.44 (0.19)
Statistical Analysis 1: Comparison: Galcanezumab vs 75 mg Rimegepant; Test type: Superiority; Mixed Models Analysis; LS Mean difference = -0.36, 95% CI 2-sided [-0.90 to 0.18]

7. Secondary Outcome: Mean Change From Baseline in the Number of Monthly Migraine Headache Days at Month 3
Description: as for outcome 5
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days per month
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 249 | 259
days per month | -5.13 (0.20) | -4.94 (0.20)
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Test type: Superiority; Mixed Models Analysis; LS Mean difference = -0.18, 95% CI 2-sided [-0.73 to 0.37]

8. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days Requiring Medication for the Acute Treatment of Migraine or Headache Across the 3-month Treatment Period.
Description: Number of monthly migraine headache days requiring medication for the acute treatment of headache is defined as the number of calendar days in a 30-day period on which migraine or probable migraine occurs and acute medication is used. Overall mean was derived from the average of month 1 through month 3. LS mean was calculated using MMRM model with treatment, month, and treatment-by-month interaction as fixed effects and baseline number of migraine headache days with acute medications use, and baseline-by-month interaction as continuous variables.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days per month
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 269 | 284
days per month | -3.95 (0.14) | -3.47 (0.13)
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Test type: Superiority; Mixed Models Analysis; LS Mean difference = -0.49, 95% CI 2-sided [-0.86 to -0.11]

9. Secondary Outcome: Mean Change From Baseline in the Migraine-Specific Quality of Life Questionnaire Version 2.1 (MSQ v2.1) at Month 3
Description: The MSQ v2.1 is a 14-item questionnaire, participant-rated scale with a 4-week recall period that measures the impact of migraine on work or daily activities, relationships with family & friends, leisure time, productivity, concentration, energy, tiredness & feelings. It consists of 14 items that address 3 domains:
  * Role Function-Restrictive (RF-R), items 1-7
  * Role Function-Preventive (RF-P), items 8-11
  * Emotional Function (EF), items 12-14
  Each item is scored from 1 (none of the time) to 6 (all of the time) and are reverse coded (value 6 to 1). Raw scores for each domain are computed as a sum of item responses, with the collective sum providing a total raw score. These were transformed to a 0-100 scale, with higher scores indicating better quality of life.
  LS mean was calculated using Analysis of covariance (ANCOVA) with main effects of treatment, the baseline number of migraine headache days category (<8 vs >=8), and the continuous fixed covariate of the baseline endpoint.
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 271 | 269
score on a scale
  Total score | 28.92 (1.07) | 24.53 (1.07)
  RF-R | 31.90 (1.20) | 26.66 (1.20)
  RF-P | 24.62 (1.02) | 20.74 (1.02)
  EF | 27.76 (1.17) | 24.58 (1.17)
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Total score; Test type: Superiority; ANCOVA; LS Mean difference = 4.39, 95% CI 2-sided [1.42 to 7.37], Standard Error of Mean 1.51
Statistical Analysis 2: Comparison: Galcanezumab vs Rimegepant; RF-R; Test type: Superiority; ANCOVA; LS Mean difference = 5.24, 95% CI 2-sided [1.90 to 8.58], Standard Error of Mean 1.70
Statistical Analysis 3: Comparison: Galcanezumab vs Rimegepant; RF-P; Test type: Superiority; ANCOVA; LS Mean difference = 3.88, 95% CI 2-sided [1.06 to 6.71], Standard Error of Mean 1.44
Statistical Analysis 4: Comparison: Galcanezumab vs Rimegepant; EF; Test type: Superiority; ANCOVA; LS Mean difference = 3.18, 95% CI 2-sided [-0.08 to 6.44], Standard Error of Mean 1.66

10. Secondary Outcome: Mean Change From Baseline on the Migraine Disability Assessment Test (MIDAS) Total Score at Month 3
Description: The MIDAS is a participant-rated scale that measures headache-related disability over a 3-month period. It consists of 5 items that measures number of days of work/school missed or days with productivity at work/school reduced to half or more; days with household work missed or days with productivity in household work reduced to half or more, and days of missed family/social/leisure activities. Each item has a numeric response range from 0 to 90 days; if days are missed from work/school or household work they are not counted as days with reduced productivity at work/school or household work. The numeric responses are summed to produce a total score ranging from 0 to 270. A higher value is indicative of more disability.
  LS mean was calculated using ANCOVA model with main effects of treatment, the baseline number of migraine headache days category (<8 vs >=8), and the continuous fixed covariate of the baseline endpoint.
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Galcanezumab | Rimegepant
Number analyzed (Participants) | 271 | 269
score on a scale | -22.54 (1.63) | -20.11 (1.63)
Statistical Analysis 1: Comparison: Galcanezumab vs Rimegepant; Test type: Superiority; ANCOVA; LS Mean difference = -2.43, 95% CI 2-sided [-6.94 to 2.08], Standard Error of Mean 2.30

ADVERSE EVENTS:
Time Frame: Baseline up to Month 3
Description: All randomized participants who received at least 1 dose of the study drug. As per the planned safety analyses, AE data was reported per treatment regimen received.
Arm/Group | Galcanezumab | Rimegepant
All-Cause Mortality (participants affected / at risk) | 0/287 | 0/293
Serious Adverse Events (participants affected / at risk) | 0/287 | 1/293
Other Adverse Events (participants affected / at risk) | 28/287 | 28/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab (N=287) | Rimegepant (N=293)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab (N=287) | Rimegepant (N=293)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 2 (2) | 4 (4)
Injection site pain (General disorders) | 2 (2) | 4 (4)
Covid-19 (Infections and infestations) | 12 (12) | 5 (5)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (6)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT05127486/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT05127486/SAP_001.pdf